CLINICAL TRIAL: NCT01689402
Title: MRI for Early Identification of Underlying Pathology in Patients With Acute Intracerebral Hemorrhage
Brief Title: MRI for the Early Evaluation of Acute Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Associate Research Professor, Consultant Neurologist, Bispebjerg Hospital
Other Study IDs: H-2-2012-009
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Hemorrhage; Intracranial Arteriovenous Malformations; Intracranial Hemorrhage, Hypertensive; Brain Neoplasms
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Arteriovenous Malformations; Intracranial Hemorrhage, Hypertensive; Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracerebral Hemorrhage Patients: Patients admitted with acute intracerebral hemorrhage within 72 hours after symptom onset.Patients are included in the study for MRI studies
  Interventions: Device: MRI Scan with the specified sequences below:

INTERVENTIONS:
Device: MRI Scan with the specified sequences below: — Standard sequences: Axial T2, axial DWI, Sagittal T1, T2 flair og axial GRE-sequence.
  Susceptibility weighted imaging (SWI)
  Chemical Shift Imaging (CSI) multivoxel spectroscopi
  Post contrast 3D box reconstruction

SUMMARY:
What happens in the borderzone of a cerebral hemorrhage remains widely onknown and furhter the best timing for doing MR to look for vascular pathology in cerebral hemorrhage has not yet been determined. In this study we do acute MRS, a non-invasive imaging mathod to detemine the biochemsty in the border zone and structural MRI for vascular malformation. We repeat structural MRI after 8 weeks.

DETAILED DESCRIPTION:
In this study we want to investigate the ability of MRI to identify underlying pathology (tumor or vascular malformations) in acute patients admitted with intracerebral hemorrhage (ICH). Today MRI-scan is normally done 3-4 weeks after symptom onset but very little is known about the early use of MRI to detect underlying pathology. This would allow an early intervension and less uncertainty for the patients.

We further want to investigate the metabolic penumbra-zone surrounding the hematoma. It is the current perception in the litterature that this zone represent a metabolic zone marked by apoptosis and inflammation rather than ischemia.

We are planning to:

When patients arrive in our stroke department they will within 7 hours be subject to MRI scan with the protocoled sequences. Standard sequences: Axial T2, axial DWI, Sagittal T1, T2 flair og axial GRE-sequence.

Susceptibility weighted imaging (SWI)

Chemical Shift Imaging (CSI) multivoxel spectroscopi

Post contrast 3D box reconstruction

After 8 weeks the patients are subject to another MRI-Scan in accordance with the standard clinical guideline to rule out underlying pathology.

After 3 month the patients are seen in the outpatient-clinic to follow-up evaluation.

To sum up the purpose of this present study is to conduct a pilot investigation of MRI in the early evaluation of ICH-patients. Second it is our intension to use multivoxel magnetic resonance spectroscopy to study the metabolic penumbra-zone surrounding the ICH.

ELIGIBILITY:
Inclusion Criteria:

* CT demonstrated ICH
* Cardiopulmonary stable
* Informed consent from patient or proxy
* No General contraindication of MRI
* Age above 18

Exclusion Criteria:

* Lack of informed consent
* lack of cooperability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with CT-demonstrated Intracerebral Hemorrhage (ICH) within 72 hours after symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
early correct diagnosis of underlying vascular malformation | 8 weeks
  Correct diagnosis based on findings on 8 weeks control MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Background] Sahni R, Weinberger J. Management of intracerebral hemorrhage. Vasc Health Risk Manag. 2007;3(5):701-9. PMID 18078021
- [Background] Delgado Almandoz JE, Schaefer PW, Goldstein JN, Rosand J, Lev MH, Gonzalez RG, Romero JM. Practical scoring system for the identification of patients with intracerebral hemorrhage at highest risk of harboring an underlying vascular etiology: the Secondary Intracerebral Hemorrhage Score. AJNR Am J Neuroradiol. 2010 Oct;31(9):1653-60. doi: 10.3174/ajnr.A2156. Epub 2010 Jun 25. PMID 20581068
- [Background] Wijman CA, Venkatasubramanian C, Bruins S, Fischbein N, Schwartz N. Utility of early MRI in the diagnosis and management of acute spontaneous intracerebral hemorrhage. Cerebrovasc Dis. 2010;30(5):456-63. doi: 10.1159/000316892. Epub 2010 Aug 24. PMID 20733299
- [Background] Diedler J, Karpel-Massler G, Sykora M, Poli S, Sakowitz OW, Veltkamp R, Steiner T. Autoregulation and brain metabolism in the perihematomal region of spontaneous intracerebral hemorrhage: an observational pilot study. J Neurol Sci. 2010 Aug 15;295(1-2):16-22. doi: 10.1016/j.jns.2010.05.027. Epub 2010 Jun 16. PMID 20557898
- [Background] Carhuapoma JR, Wang PY, Beauchamp NJ, Keyl PM, Hanley DF, Barker PB. Diffusion-weighted MRI and proton MR spectroscopic imaging in the study of secondary neuronal injury after intracerebral hemorrhage. Stroke. 2000 Mar;31(3):726-32. doi: 10.1161/01.str.31.3.726. PMID 10700511
- [Background] Carhuapoma JR, Wang P, Beauchamp NJ, Hanley DF, Barker PB. Diffusion-perfusion MR evaluation and spectroscopy before and after surgical therapy for intracerebral hemorrhage. Neurocrit Care. 2005;2(1):23-7. doi: 10.1385/NCC:2:1:023. PMID 16174964
- [Background] Karaszewski B, Thomas RG, Chappell FM, Armitage PA, Carpenter TK, Lymer GK, Dennis MS, Marshall I, Wardlaw JM. Brain choline concentration. Early quantitative marker of ischemia and infarct expansion? Neurology. 2010 Sep 7;75(10):850-6. doi: 10.1212/WNL.0b013e3181f11bf1. PMID 20819997